CLINICAL TRIAL: NCT00001164
Title: Studies of Patients With Skin Disease, Patients With Neurological Degenerations, and Normal Volunteers
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 780099; 78-C-0099
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-05 (Estimated); Status verified 2000-06

CONDITIONS: Healthy; Muscular Dystrophy; Retinal Degeneration; Skin Diseases; Virus Diseases
Keywords: Genetic Evaluation; Immunologic Evaluations; Inflammatory Skin Disease; Muscular Dystrophies; Neoplastic Skin Diseases; Neuronal Degenerations; Retinal Degenerations; Viral Diseases
MeSH Terms: conditions — Muscular Dystrophies; Retinal Degeneration; Skin Diseases; Virus Diseases; Dermatitis

SUMMARY:
It is proposed that patients with skin disease due to presumed immunologic, genetic or viral-induced abnormalities, patients with neurological degenerations, and normal controls be evaluated with various in vitro studies of immunologic, genetic, and virologic function. This is to include studies of peripheral blood (cells and serum) as well as studies of skin obtained with a biopsy instrument. In addition, studies of gastrointestinal function will be performed where appropriate.

DETAILED DESCRIPTION:
It is proposed that patients with skin disease due to presumed immunologic, genetic or viral-induced abnormalities, patients with neurological degenerations, and normal controls be evaluated with various in vitro studies of immunologic, genetic, and virologic function. This is to include studies of peripheral blood (cells and serum) as well as studies of skin obtained with a biopsy instrument. In addition, studies of gastrointestinal function will be performed where appropriate.

ELIGIBILITY:
Patients with skin diseases of presumed genetic, immunologic, or virologic origin are eligible.

Patients with neurological degenerations are eligible, including patients with inflammatory, neoplastic and viral skin diseases and also heterozygous carriers of such inherited diseases.

Volunteers without skin diseases are eligible, except children.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Dates: Start 1978-07; Study Completion 2000-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Kraemer KH, Coon HG, Petinga RA, Barrett SF, Rahe AE, Robbins JH. Genetic heterogeneity in xeroderma pigmentosum: complementation groups and their relationship to DNA repair rates. Proc Natl Acad Sci U S A. 1975 Jan;72(1):59-63. doi: 10.1073/pnas.72.1.59. PMID 164028
- [Background] Yaoita H, Katz SI. Immunoelectronmicroscopic localization of IgA in skin of patients with dermatitis herpetiformis. J Invest Dermatol. 1976 Oct;67(4):502-6. doi: 10.1111/1523-1747.ep12664534. PMID 972257